CLINICAL TRIAL: NCT02450968
Title: Dexamethasone for Prophylaxis of Acute Mountain Sickness in Patients With Chronic Obstructive Pulmonary Disease Travelling to Altitude
Brief Title: Altitude Related Illness In Patients With Respiratory Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EK15-2015
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: airway disease; bronchitis; emphysema; lung; treatment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 4 mg capsules, twice per day, orally
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo capsules twice per day, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Dexamethasone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Randomized, placebo controlled trial evaluating efficacy of dexamethasone in preventing acute mountain sickness in lowlanders with chronic obstructive lung disease travelling from 700 m to 3200 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the efficacy of dexamethasone prophylaxis in reducing the incidence of acute mountain sickness in lowlanders with chronic obstructive pulmonary disease travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (700m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3200 m), and stay there for 2 days. Dexamethasone 2x4mg/day (or placebo), will be administered before departure at 700 m and during the stay at altitude. Outcomes will be assessed during the stay at 3200 m.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease (COPD), GOLD grade 1-2
* Living at low altitude (<800m)

Exclusion Criteria:

* COPD exacerbation
* severe COPD, GOLD grade 3 or 4
* arterial oxygen saturation <92% at low altitude (<800 m)
* Diabetes, uncontrolled cardiovascular disease such as systemic arterial hypertension, coronary artery disease; previous stroke; pneumothorax in the last 2 months, untreated or symptomatic peptic ulcer disease, glaucoma, obstructive sleep apnea.
* Internal, neurologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day).
* pregnant or nursing patients

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Acute mountain sickness, cumulative incidence | day 3 at 3200 m
  Difference between dexamethasone and placebo group in cumulative incidence of acute mountain sickness assessed by the environmental symptoms questionnaire cerebral subscale (score >=0.7)

SECONDARY OUTCOMES:
Severe hypoxemia | day 1 to 3 at 3200m
  Number of participants in the dexamethasone and placebo group with arterial oxygen saturation measured by pulse oximetry less than 75% for more than 30 min or less than 70% for more than 15 min.
Acute mountain sickness, severity | day 1, day 2, day 3 at 3200 m
  Difference between dexamethasone and placebo group in the acute mountain sickness severity assessed by the environmental symptoms questionnaire cerebral subscale
6 min walk distance | Day 2 at 3200 m
  Difference in the distance walked in 6 min between the dexamethasone and placebo group
Perceived exertion | Day 2 at 3200 m
  Difference in the perceived exertion rated with the Borg CR10 scale between the dexamethasone and placebo group
Spirometry | Day 2 at 3200 m
  Difference in the spirometric variables between the dexamethasone and placebo group
Arterial blood gases | Day 2 at 3200 m
  Difference in arterial oxygen partial pressure, carbon dioxide partial pressure, and pH between the dexamethasone and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

REFERENCES:
- [Derived] Preiss H, Mayer L, Furian M, Schneider SR, Muller J, Saxer S, Mademilov M, Titz A, Shehab A, Reimann L, Sooronbaev T, Tanner FC, Bloch KE, Ulrich S, Lichtblau M. Right ventricular strain impairment due to hypoxia in patients with COPD: a post hoc analysis of two randomised controlled trials. Open Heart. 2025 Jan 4;12(1):e002837. doi: 10.1136/openhrt-2024-002837. PMID 39756820
- [Derived] Muralt L, Furian M, Lichtblau M, Aeschbacher SS, Clark RA, Estebesova B, Sheraliev U, Marazhapov N, Osmonov B, Bisang M, Ulrich S, Latshang TD, Ulrich S, Sooronbaev TM, Bloch KE. Postural Control in Lowlanders With COPD Traveling to 3100 m: Data From a Randomized Trial Evaluating the Effect of Preventive Dexamethasone Treatment. Front Physiol. 2018 Jun 22;9:752. doi: 10.3389/fphys.2018.00752. eCollection 2018. PMID 29988503
- [Derived] Furian M, Lichtblau M, Aeschbacher SS, Estebesova B, Emilov B, Sheraliev U, Marazhapov NH, Mademilov M, Osmonov B, Bisang M, Ulrich S, Latshang TD, Ulrich S, Sooronbaev TM, Bloch KE. Efficacy of Dexamethasone in Preventing Acute Mountain Sickness in COPD Patients: Randomized Trial. Chest. 2018 Oct;154(4):788-797. doi: 10.1016/j.chest.2018.06.006. Epub 2018 Jul 10. PMID 29909285